CLINICAL TRIAL: NCT06120816
Title: Phase 1 Single Centre, Open-labeled Clinical Trial to Evaluate the Safety and Tolerability of Topical Nitric Oxide Releasing Mouthwash (NORM) for the Management of Oropharyngeal Candidiasis
Brief Title: Nitric Oxide Releasing Mouthwash (NORM) for the Management of Oropharyngeal Candidiasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanotize Research and Development corp. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NORM-POC-01
Record Dates: First submitted 2023-11-01; First posted 2023-11-07 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Candidiasis, Oral
Keywords: oral candidiasis
MeSH Terms: conditions — Candidiasis, Oral | interventions — Nitric Oxide

STUDY DESIGN:
Intervention Model Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nitric Oxide Releasing Mouthwash (Experimental): Nitric Oxide Releasing Mouthwash (NORM) liquid producing NO at 266 ppm*min in 20mL
  Interventions: Drug: Nitric Oxide

INTERVENTIONS:
Drug: Nitric Oxide — Nitric Oxide Releasing Mouthwash will be self-administered by the participant three times throughout the day for 21 days. The intervention solution will be poured into their mouth from a medication cup containing 20 mL of the solution. Total exposure to study intervention will be a maximum of 63 treatments totaling 1,260 mL. All participants will be monitored for 7 days post-last treatment dose (to Day 28).
  Other Names: Nitric Oxide Releasing Mouthwash

SUMMARY:
Phase 1 Single Centre, open-labeled Clinical Trial to Evaluate the Safety and Tolerability of Topical Nitric Oxide Releasing Mouthwash (NORM) for the Management of Oropharyngeal Candidiasis.

Participants that meet all inclusion and exclusion criteria will be enrolled to receive open label NORM 3 doses/day for three weeks.

DETAILED DESCRIPTION:
This is a single-center, open-label phase 1 clinical trial to evaluate NORM safety, tolerance and ability to eliminate Candida sp from the oropharyngeal cavity.

Adult volunteer patients with dry mouth and confirmed presence of candida (by oral smear due to any cause will be eligible, including autoimmune disease, idiopathic (aging, tobacco, approved inhaled recreational drug, or alcohol use), and medical management including chemotherapy-induced, radiotherapy-induced, bone marrow transplantation-induced, medication use including antibiotics, anti-inflammatories, etc.

Sufficient participants will be enrolled to achieve 10 evaluable participants. Participants who are currently pursuing other forms of treatment (within 2 weeks prior to enrollment) will be excluded from the study (unless participant agrees to a two weeks wash out period).

ELIGIBILITY:
Inclusion Criteria:

1. At least 19 years old at the time of consent.
2. Participants must be diagnosed with clinical candidiasis.
3. Have no acute illnesses or hospitalizations within 30 days prior to enrollment, no planned procedures during the anticipated study participation, and no newly diagnosed chronic illnesses that are not deemed stable by the participant's primary care physician), in the opinion of the Investigator, based on medical history (i.e., absence of any clinically relevant abnormality) during Screening.
4. Participants must not have been part of any clinical trial for the past 30 days and may not be taking any other investigational therapy related to treatment of candidiasis.
5. If female, be surgically sterile or post-menopausal (no menses for at least 12 months), or if of childbearing potential, must be using an acceptable method of contraception such as a combination estrogen/progestin hormonal contraceptive (oral or injected) for at least 1 month prior to Day -14, or such items as an intrauterine device (IUD), intrauterine system (IUS), transdermal hormonal implant, vaginal hormonal ring, or 2 forms of the following: diaphragm, cervical cap, patch, condom, spermicide, or sponge. Total abstinence is permitted. If local regulations deviate from the previously listed contraception methods to prevent pregnancy, local requirements will apply. In addition, females of childbearing potential must agree to continue to use their method of birth control for the duration of the study.
6. If male, be surgically sterile, or agree to use appropriate contraception (latex condom with spermicide) when engaging in sexual activity and agree to not donate sperm for the duration of the study.
7. Be able to understand and provide written, informed consent.
8. Must be willing and able to manage a treatment regimen and attend assessment study visits.

Exclusion Criteria:

1. Participants with mucosal/oral ulceration
2. No prior antifungal therapies for a minimum 2-week prior to enrollment
3. Participants with other conditions considered by the investigator to be reasons for disqualification that may jeopardize patient safety or interfere with the objectives of the trial (e.g., acute illness or exacerbation of chronic illness, lack of motivation, history of poor compliance, neurologically or mentally disabled)
4. Females who are breastfeeding, pregnant, or attempting to become pregnant.
5. Participants with hypersensitivity to any of the product's ingredients.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2024-01-20 (Actual); Primary Completion 2024-05-25 (Actual); Study Completion 2024-05-25 (Actual)

PRIMARY OUTCOMES:
To assess the tolerability of NORM in participants with candidiasis. | 21 days
  Intolerance (i.e., oral cavity, dental, and/or lingual irritation or sensitivity (pain, swelling, erythema, discharge)), dysgeusia, or discoloration of oral cavity/teeth/tongue) as assessed by number of patients that terminate NORM treatment.

SECONDARY OUTCOMES:
To assess the effectiveness of NORM to resolve oral fungal infection | 21 days
  Assess the number of participants who experience clearing of the infection by negative smear/culture
To assess the effectiveness of NORM to resolve clinical symptoms of candidiasis | 21 days
  Mean time to achieve clearing of clinical infection (no symptoms [0] or mild [1]) from Baseline until Day 21
To assess the effectiveness of NORM to reduce the need for an oral antifungal agent | 21 days
  Proportion of participants that require nystatin intervention

OTHER OUTCOMES:
To categorize the major reasons impacting the tolerance of NORM during oral administration | 21 days
  Tolerance as assessed by number of patient reported outcomes (PRO) of irritation and dysgeusia of the rinse, dental sensitivity while willing to continue to use the rinse
Determine incidence and severity of adverse reactions | 21 days
  Safety as assessed by number and severity of adverse events
To assess reoccurrence of candidiasis | 28 days
  Proportion of participants with reemergence of candidiasis infection
To assess of exacerbation of candidiasis | 28 days
  Proportion of participants with an increased Candida sp. associated with their lesions (determined as an increase of 2 or more semi-quantitative steps (e.g., scant to moderate or light to heavy))

CONTACTS AND LOCATIONS:
Overall Officials: Keith Moore, PHARMMD, Study Director — SaNOtize R&D Corp; Joel Epstein, Principal Investigator — Atlantis Dental Cambie
Locations (1):
- Atlantis Dental Cambie, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://wartsstudy.ca